CLINICAL TRIAL: NCT02274922
Title: Evaluation of Immunochromatographic Tests for Campylobacter Detection in Stools
Acronym: CAMPYTEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/05
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Gastroenteritis
Keywords: Campylobacter diagnosis,; immuno-chromatographic test, ELISA, PCR, culture, stool; ELISA,; PCR,; culture, stool
MeSH Terms: conditions — Gastroenteritis; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serology control
Oversight: Data Monitoring Committee: No

SUMMARY:
For a long time, culture was the only way to detect Campylobacter. It appears that rapid immunochromatographic tests (ICT) have detected more positive cases compared to culture, ELISA and molecular tests. The aim of our study is to evaluate the specificity of the ICT which are really interesting tools to use since they allow a diagnosis in about 15 min, in comparison to different methods of detection even serology.

DETAILED DESCRIPTION:
All of the patients coming to an emergency care unit and for whom a stool culture is prescribed will be included, corresponding to an estimate number of 1,000 patients for two years. Every stools will be tested for Campylobacter using two different ICT tests in addition to the standard culture. Then, in function of the ICT test result : 1) in case of negative result, no other Campylobacter detection will be performed except the standard culture, 2) in case of positive result, stools will be tested for Campylobacter by two ELISA tests, one PCR and a serology at two different times (D0 and D15) will be performed. Around 70 patients should be detected positive with ICTs, according to precedent studies. The 70 patients detected positive with at least one of the two ICT will have a serology control 15 days after the ICT test. The reference test will be the combination of culture result, evolution of the serology between D0 and D15 and the PCR and ELISA results. We want to define a procedure to follow in order to detect as soon as possible and with the best results, the Campylobacters in the stool of patients. This has the aim of being able to manage patients who need appropriate antibiotic treatment, and also to reduce the time of hospitalization of patients quickly detected as suffering from a Campylobacter infection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient of any age (pediatric and adult) and any sex
* Admitted to the emergency hospital for less than 48 who had a stool sample for stool culture including women and elderly patients over 65 years

Exclusion Criteria:

* there is no " non-inclusion " criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the patients coming to an emergency care unit and for whom a stool culture is prescribed will be included, corresponding to an estimate number of 1,000 patients for two years.
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
positive Campylobacter detection with ICT | The day of inclusion

SECONDARY OUTCOMES:
result of PCR | The day of inclusion
result of PCR | 15 days after inclusion
stool culture | The day of inclusion
stool culture | 15 days after inclusion
ELISA | The day of inclusion
ELISA | 15 days after inclusion
serology for Campylobacter detection | The day of inclusion
serology for Campylobacter detection | 15 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Perez Paul, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique du CHU de Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France